CLINICAL TRIAL: NCT04708756
Title: Collabree: A Targeted Behavioral Economics-based Intervention to Improve Medication Adherence in Patients With Hypertension
Brief Title: Collabree: An Intervention to Improve the Regularity of Medication Intake
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Collabree AG (Industry)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COLLABREE-S
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Hypertension; Medication Adherence
Keywords: Digital Health; Behavioral Change
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group A (Experimental): Patients receive the Collabree mobile phone application with a specific set of functions and standard care.
  Interventions: Behavioral: Collabree Mobile Phone Application Medication Adherence Booster
- Intervention Group B (Experimental): Patients receive the Collabree mobile phone application with a specific set of functions and standard care.
  Interventions: Behavioral: Collabree Mobile Phone Application Medication Adherence Booster (simplified version)
- Control Group (No Intervention): Patients will not receive the Collabree application and will continue to receive standard care.

INTERVENTIONS:
Behavioral: Collabree Mobile Phone Application Medication Adherence Booster (simplified version) — Patients take part in a 90-day program to promote medication adherence and a 90-day follow-up through the Collabree application. Patients will receive more information as to the exact functions and use of the mobile phone application when the application is installed on their mobile phone. Patients will receive standard care.
  Arms: Intervention Group B
Behavioral: Collabree Mobile Phone Application Medication Adherence Booster — Patients take part in a 90-day program to promote medication adherence and a 90-day follow-up through the Collabree application. Patients will receive more information as to the exact functions and use of the mobile phone application when the application is installed on their mobile phone. Patients will receive standard care.
  Arms: Intervention Group A

SUMMARY:
This a clinical study to improve medication adherence among patients with hypertension in Switzerland. Adult men and women who suffer from high blood pressure and have been prescribed a therapy consisting of at least 4 tablets per day can participate in this study.

The investigators intend to examine whether Collabree, a mobile phone application, is effective in supporting patients with hypertension to more successfully following their therapy plan. The study will also investigate if the use of Collabree can help lower blood pressure.

The study consists of 4 visits that take place during a 90-day adherence promotion program plus a 90-day follow-up period. There is also a screening visit before the study to determine whether the participants qualify for the study. The visits are carried out at the University Hospital Basel. Each visit lasts about 1-2 hours. During the visits, blood pressure is measured in the clinic and also through 24-hour ambulatory blood pressure monitoring (ABPM). Participants will also fill out questionnaires.

Participants are randomly assigned to one of 3 groups in a ratio of 1: 1: 1. Two of these groups will receive the Collabree mobile phone application. All participants will receive a box for storing their antihypertensive medication. This box serves as a system for measuring medication intake as it records the time the box is opened and closed. Standard care will given to all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent as documented by signature
2. Over 18 years of age at date of randomization
3. Primary or secondary arterial hypertension
4. Patient in an outpatient clinical setting
5. Prescribed a therapy consisting of 4 or more tablets taken per day
6. Stable medication regime that patient has been taking for at least 4 weeks
7. Participant administers their own medications
8. Participant owns a smartphone with a data plan or constant internet access during the study visits and at home to use the application
9. Minimal required smartphone operating system is iOS 12 and Android 8 (Oreo)
10. Adequate communication in German or Swiss-German (all study documentation will only be set to the German language).

Exclusion Criteria:

1. Cognitive impairment that limits ability to understand and complete questionnaires
2. Ongoing evaluation for secondary forms of hypertension
3. 3. Changes in the participant's medication treatment plan after the baseline visit during the intervention period, unless due to a diagnosis of symptomatic hypotension (in-clinic blood pressure below 110/60 mmHg and symptoms of orthostasis or dizziness) or stage 2 hypertension (in-clinic blood pressure > 160/100 mmHg); after the endpoint (day 90) visit, a change in the treatment plan will be permitted
4. Uncontrolled hypertension (in-clinic blood pressure > 180/110 mmHg)
5. Inability to operate a mobile phone and the Collabree application
6. Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
7. Pregnancy or intention to become pregnant in next 6 months
8. Enrollment of the Sponsor or Investigator, their family members, employees and other dependent persons
9. Participation in another clinical trial
10. Physician-estimated life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | 90 days
  Difference between intervention Group A and the control group in mean medication adherence at endpoint (i.e. the endpoint visit at 90 days) as measured by medication events.

SECONDARY OUTCOMES:
Medication adherence (3 group comparison) | 90 days
  Mean change from baseline in medication adherence (monitored by medication events) at endpoint for the intervention Group A vs. intervention Group B relative to the control group.
Self-reported medication adherence | 90 days
  Mean change from baseline in in-app medication adherence (defined as the number of medications self-reported as "taken" during the intervention period of 90 days divided by the number of prescribed medications listed in the in-app medication plan in that same time period) at endpoint for the intervention Group A vs. intervention Group B relative to the control group.
Self-assessed medication adherence | 90 days
  Mean change from baseline in the score on the Hill-Bone Scale (German version) questionnaire on medication adherence for the intervention Group A vs. intervention Group B relative to the control group at endpoint.
Blood pressure | 180 days
  Linear change in systolic and diastolic blood pressure (24h ABPM and in-clinic blood pressure measurement) across time from baseline to follow-up as assessed with a linear mixed regression model. This linear change will then be compared for the intervention Group A and intervention Group B relative to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Burkard, MD, ISHF, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided